CLINICAL TRIAL: NCT00637689
Title: Improving Outcomes Assessment in Chronic GVHD
Status: Active, not recruiting | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of Minnesota (Other); Stanford University (Other); Dana-Farber Cancer Institute (Other); Vanderbilt University (Other); Medical College of Wisconsin (Other); Washington University School of Medicine (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); Memorial Sloan Kettering Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: FHCRC-2192.00; U01CA118953-01A1 (NIH); IR-6531 (Other: FHCRC); RG1000709 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: Chronic graft versus host disease; Allogeneic hematopoietic cell transplantation; Biomarkers; Response criteria; Surrogate endpoints; Natural history
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Some centers are collecting serum, plasma, cells and urine.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to see if recent guidelines proposed by the National Institutes of Health for the diagnosis, staging, and response assessment of people with chronic GVHD can improve our understanding of this complication. We will accomplish our goals by studying a large number of people with chronic GVHD over several years using information collected from health care providers, patients, laboratory studies and diagnostic tests. Several transplant centers in the United States are collaborating on this project.

DETAILED DESCRIPTION:
Chronic graft-versus-host disease (GVHD) is one of the most devastating long-term complications after infusion of allogeneic hematopoietic stem cells, and it remains one of the major barriers to successful transplantation. Relatively little progress has been made in understanding and improving treatments for chronic GVHD over the last 20 years, and the survival rate after diagnosis of chronic GVHD has barely improved despite advances in supportive care. The National Institutes of Health convened a Consensus Conference on this topic in June 2004 and recently published its recommendations on improving research methods in a series of six papers.

In our study, we will establish a multi-center, observational, longitudinal cohort in order to improve outcomes assessment in chronic GVHD with the specific aims of (1) validating prognostic factors for risk stratification; and (2) defining significant variables for a chronic GVHD activity index that predicts short-term (provider perception of change, patient perception of change, and changes in immunosuppressive medications) and longer-term outcomes (overall survival, time to discontinuation of systemic immunosuppressive therapy, and functional impairments). This goal will be accomplished by assembling a large modern cohort of people with chronic GVHD at four large core transplant centers. Approximately 700 people (half prevalent cases, half incident cases) with chronic GVHD will be enrolled. Every 3-6 months we will collect both objective and subjective measures reflecting disease activity, response to therapy, detailed physician assessments about organ involvement, and patient self-assessments about symptoms, functional status, and quality of life. Data will be used to test published hypotheses and the new recommendations emanating from the NIH Consensus conference. We will also be able to provide the detailed data needed to understand modern trends in chronic GVHD incidence, manifestations, and response to treatment. These studies are needed to operationalize the recommendations of the NIH Consensus conference, advance our understanding of chronic GVHD, and enhance our ability to conduct clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 2 years
* Prior allogeneic stem cell transplant, with any graft source, donor type, and GVHD prophylaxis allowed
* Clinical or histologic diagnosis of chronic GVHD (overlap syndrome with acute GVHD is allowed
* Need for systemic treatment, defined as any medication or intervention delivered systemically, including extracorporeal photopheresis. If a patient only received topical or local therapy at diagnosis, but subsequently requires systemic treatment, they may be enrolled upon initiation of systemic therapy. (Note, these patients will be classified as incident or prevalent cases depending on time from chronic GVHD diagnosis, not start of systemic therapy)
* If a prevalent case (defined as enrollment three or more months after chronic GVHD diagnosis), then subject must be within 2 years of stem cell infusion
* If an incident case (enrollment less than 3 months after chronic GVHD diagnosis) then no limitation on time from transplantation
* No evidence of primary disease relapseProgression-free for their malignancy at enrollment (no evidence of primary disease progression since transplant, although residual disease may still be present)
* Evaluation at the transplant center at the time of study enrollment
* Signed, informed consent and if applicable, child assent

Exclusion Criteria:

* Inability to comply with study procedures
* Anticipated survival less than 6 months due to co-morbid disease

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with chronic GVHD
Sampling Method: Non-Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
Time to discontinuation of immunosuppression | 3 years
Functional impairments | 3 years

SECONDARY OUTCOMES:
Provider perception of change | 6 months
Patient perception of change | 6 months
Changes in immunosuppressive medications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J Lee, MD MPH, Principal Investigator — Fred Hutchinson Cancer Center
Locations (9):
- United States (9):
  - Stanford University, Stanford, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering, New York, New York
  - Vanderbilt University, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Inamoto Y, Martin PJ, Onstad LE, Cheng GS, Williams KM, Pusic I, Ho VT, Arora M, Pidala J, Flowers MED, Gooley TA, Lawler RL, Hansen JA, Lee SJ. Relevance of Plasma Matrix Metalloproteinase-9 for Bronchiolitis Obliterans Syndrome after Allogeneic Hematopoietic Cell Transplantation. Transplant Cell Ther. 2021 Sep;27(9):759.e1-759.e8. doi: 10.1016/j.jtct.2021.06.006. Epub 2021 Jun 12. PMID 34126278
- [Derived] Gandelman JS, Byrne MT, Mistry AM, Polikowsky HG, Diggins KE, Chen H, Lee SJ, Arora M, Cutler C, Flowers M, Pidala J, Irish JM, Jagasia MH. Machine learning reveals chronic graft-versus-host disease phenotypes and stratifies survival after stem cell transplant for hematologic malignancies. Haematologica. 2019 Jan;104(1):189-196. doi: 10.3324/haematol.2018.193441. Epub 2018 Sep 20. PMID 30237265
- [Derived] Martin PJ, Storer BE, Inamoto Y, Flowers MED, Carpenter PA, Pidala J, Palmer J, Arora M, Jagasia M, Arai S, Cutler CS, Lee SJ. An endpoint associated with clinical benefit after initial treatment of chronic graft-versus-host disease. Blood. 2017 Jul 20;130(3):360-367. doi: 10.1182/blood-2017-03-775767. Epub 2017 May 11. PMID 28495794
- [Derived] Palmer J, Chai X, Pidala J, Inamoto Y, Martin PJ, Storer B, Pusic I, Flowers ME, Arora M, Pavletic SZ, Lee SJ. Predictors of survival, nonrelapse mortality, and failure-free survival in patients treated for chronic graft-versus-host disease. Blood. 2016 Jan 7;127(1):160-6. doi: 10.1182/blood-2015-08-662874. Epub 2015 Nov 2. PMID 26527676
- [Derived] Palmer J, Chai X, Martin PJ, Weisdorf D, Inamoto Y, Pidala J, Jagasia M, Pavletic S, Cutler C, Vogelsang G, Arai S, Flowers ME, Lee SJ. Failure-free survival in a prospective cohort of patients with chronic graft-versus-host disease. Haematologica. 2015 May;100(5):690-5. doi: 10.3324/haematol.2014.117283. Epub 2015 Feb 24. PMID 25715403
- [Derived] Treister N, Chai X, Kurland B, Pavletic S, Weisdorf D, Pidala J, Palmer J, Martin P, Inamoto Y, Arora M, Flowers M, Jacobsohn D, Jagasia M, Arai S, Lee SJ, Cutler C. Measurement of oral chronic GVHD: results from the Chronic GVHD Consortium. Bone Marrow Transplant. 2013 Aug;48(8):1123-8. doi: 10.1038/bmt.2012.285. Epub 2013 Jan 28. PMID 23353804
- [Derived] Arai S, Jagasia M, Storer B, Chai X, Pidala J, Cutler C, Arora M, Weisdorf DJ, Flowers ME, Martin PJ, Palmer J, Jacobsohn D, Pavletic SZ, Vogelsang GB, Lee SJ. Global and organ-specific chronic graft-versus-host disease severity according to the 2005 NIH Consensus Criteria. Blood. 2011 Oct 13;118(15):4242-9. doi: 10.1182/blood-2011-03-344390. Epub 2011 Jul 26. PMID 21791424